**NCT number** :123436

**Document date: 20.12.2022** 

EVALUATION OF THE EFFECT OF MOBILE APPLICATION BASED WOUND HEALING PROCESS COURSE ON CLINICAL REASONING SKILLS OF NURSING STUDENTS

**SUMMARY** 

Today, there is a need to integrate rapidly developing technology into educational environments and to structure educational environments. Micro-learning modules have been used in e-learning platforms recently, with short content and user focus. This randomized controlled study was planned to evaluation the effect of mobile application-based wound healing course on clinical reasoning skills of nursing students. The population of the study will consist of students enrolled in the Surgical Diseases Nursing course in the fall and springs semester of the 2022-2023 academic year in the Department of Nursing at the Faculty of Health Sciences of Karadeniz Technical University. The students enrolled in the Surgical Diseases Nursing course in the fall semester will form the control group, while the students enrolled in the spring semester will form the experimental group. Students in the control group will take the wound healing process course with the presentation of the trainer, and the students in the experimental group will take micro-learning courses. Data will be collected with the "Student Information Form", "Wound Healing Process Information Form" and "Micro-Learning Based Mobile Application Evaluation Form". In addition, students will be evaluated on the simulator of clinical decision-making processes. The micro-learning course will remain open to students in the experimental group for 31 day. In order to measure the permanence of the knowledge, the "Wound Healing Process Information Form" will be filled in again after 31 days to the students in the control and experimental groups in line with the literature. In addition, students will be evaluated on the simulator of clinical decision-making processes. The results obtained after the application will be analyzed and the effect of the micro-learning course on the decision-making processes of the students will be determined.

Keywords: Education, Nursing, Student, Learning, Wound healing